CLINICAL TRIAL: NCT02979262
Title: IPV and Fatherhood Intervention in Residential Substance Abuse Treatment
Brief Title: Intimate Partner Violence and Fatherhood Intervention in Residential Substance Abuse Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34DA038763-01A1 (NIH); 1R34DA038763-01A1 (NIH)
Record Dates: First submitted 2016-10-04; First posted 2016-12-01 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2016-11

CONDITIONS: Intimate Partner Violence; Substance Abuse/Addiction; Child Maltreatment
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fathers for Change (Experimental): Fathers for Change treatment begins with individual-focused sessions followed by co-parenting focused sessions and ending with restorative parenting sessions. The areas of focus for each of the three phases of Fathers for Change are: 1) abstinence from SA and violence; 2) co-parenting; 3) parenting/father-child relationship. Treatment begins with motivational enhancement by focusing the role of men as fathers to their young children, child development and the impact of violence and SA on parenting, and the father's own childhood experiences of SA and violence to highlight the multigenerational nature of these problems. The program then focuses on skills training in the following areas: reducing automatic hostile cognitions and increasing emotion regulation skills, 2) communication and problem solving around co-parenting, and 3) restorative parenting.
  Interventions: Behavioral: Fathers for Change
- Parent Education (PE) (Active Comparator): PE is an individual intervention.PE was developed to represent parent education and support that is typically available to parents with substance use problems who are at high risk for neglecting their children. Fathers enrolled in PE will meet weekly for one hour with a PE counselor who will provide assistance in solving problems related to family basic needs (e.g., health care, child care, housing and education). The PE counselor will provide a choice of pamphlets on age-related parenting topics each week from a series of pamphlets designed for work with substance abusing parents. Sample pamphlet topics include routines and rituals, ages and milestones, alternatives to spanking, and nutrition and fitness.
  Interventions: Behavioral: Parent Education

INTERVENTIONS:
Behavioral: Fathers for Change
  Arms: Fathers for Change
Behavioral: Parent Education
  Arms: Parent Education (PE)

SUMMARY:
The proposed stage 1 intervention development study is designed to address two significant co-occurring issues for fathers with substance abuse (SA) problems: Intimate partner violence (IPV) and child maltreatment (CM). SA treatment programs are an important avenue to reduce family violence because SA treatment alone does not result in an end to these behaviors. Currently available interventions have had little success in reducing male IPV. Fathers for Change, an integrated outpatient intervention, shows promise as an intervention model targeting the intersection of SA, IPV, and CM. The intervention uses men's roles as fathers as a motivation for change and targets factors that are known to trigger SA, IPV and CM: hostile cognitions and poor emotion regulation. An intervention of this sort has not been integrated and tested as part of a residential substance abuse program for men. This project is a pilot study of 60 fathers randomly assigned to Fathers for Change or a Parent Education Program (PE) comparison. The initial feasibility of the Fathers for Change will be assessed by comparing it to PE in the areas of: participant completion rates, hostile cognitions, emotion regulation, SA relapse, IPV, and CM risk behaviors (negative parenting). Change in hostile cognitions and emotion regulation will be examined as the mechanisms through which Fathers for Change reduces relapse, IPV and CM risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. meet current DSM-5 criteria for substance use disorder of alcohol, cocaine, marijuana, amphetamines, or opiates at the time of admission to Westcare; (2) report physical violence in an intimate relationship (pushing, slapping, kicking) within 6 months of admission to the program (based on court/police records or self- report); and (3) have at least one biological child under the age of 12 with whom they lived or had at least once per month visitation prior to admission to Westcare. Each will agree to have their female co-parents contacted for participation as collateral informants and will provide the contact information. If a participant has more than one child in the age range, the youngest child will be the target of assessment. Female co-parents (the target children's mothers) will be invited to participate as collateral informants on research assessments and to participate in a portion (2 -4) of the intervention sessions. If a female co-parent does not consent to participate, a male participant will still be allowed to enroll in the study if he meets eligibility criteria

Exclusion Criteria:

* Individuals will be excluded who: 1) Have histories of severe physical violence (e.g. strangulation, causing hospitalization) based on police records, self or partner reports; 2) Men who have an active FULL/NO CONTACT protective order pertaining to their partner or child (Westcare has access to criminal record/court information for all of it's residential clients. Participants will sign releases of information during informed consent to allow the study team to access this information to determine eligibility); 3) Have cognitive impairment (a mini mental state score <25); 4) Have major medical complications such as a head injury or HIV dementia that may also be a confound in the study interventions; 5) Have current untreated psychotic or bipolar disorder (reported by history, as part of the Westcare record, or self-report); or 6) Are currently suicidal or homicidal. If potential participants have a prior diagnosis of bipolar or psychotic disorder that is currently treated and symptoms are well managed based on initial study interview and after collateral contact with the Westcare treatment team, they may participate in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Westcare Inc. Davis Bradley Building, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fathers were recruited from two 6-month men's residential substance use treatment facilities. Both programs followed a 12-step facilitation therapeutic milieu approach. Information about the study was provided by facility staff to men who entered the facility, completed 30 days of treatment and had a biological child under the age of 16.
Pre-assignment Details: Screening: 1) had some contact with his children via phone, letters or in person visits; 2) reported either physical or psychological aggression toward his female co-parent in the last 12 months; and 3) could complete study interviews and intervention in English. Eligible men met individually with an RA to complete baseline measures.
Groups:
- Fathers for Change: Fathers for Change treatment begins with individual-focused sessions followed by co-parenting focused sessions and ending with restorative parenting sessions. The areas of focus for each of the three phases of Fathers for Change are: 1) abstinence from SA and violence; 2) co-parenting; 3) parenting/father-child relationship. Treatment begins with motivational enhancement by focusing the role of men as fathers to their young children, child development and the impact of violence and SA on parenting, and the father's own childhood experiences of SA and violence to highlight the multigenerational nature of these problems. The program then focuses on skills training in the following areas: reducing automatic hostile cognitions and increasing emotion regulation skills, 2) communication and problem solving around co-parenting, and 3) restorative parenting.
  Fathers for Change
- Parent Education (PE): PE is an individual intervention.PE was developed to represent parent education and support that is typically available to parents with substance use problems who are at high risk for neglecting their children. Fathers enrolled in PE will meet weekly for one hour with a PE counselor who will provide assistance in solving problems related to family basic needs (e.g., health care, child care, housing and education). The PE counselor will provide a choice of pamphlets on age-related parenting topics each week from a series of pamphlets designed for work with substance abusing parents. Sample pamphlet topics include routines and rituals, ages and milestones, alternatives to spanking, and nutrition and fitness.
  Parent Education
Period: Overall Study
Arm/Group | Fathers for Change | Parent Education (PE)
Started | 33 | 29
Received Allocated Intervention | 30 | 27
Completed | 21 | 20
Not Completed | 12 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fathers for Change | Parent Education (PE) | Total
Number analyzed (Participants) | 33 | 29 | 62
Age, Continuous [Mean (Standard Deviation); unit: year] | 36.82 (9.07) | 34.76 (6.28) | 35.85 (7.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 33 | 29 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic Minority | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 33 | 29 | 62
Child Abuse History [Count of Participants; unit: Participants]
  Physical Abuse History | 6 | 8 | 14
  Sexual Abuse History | 4 | 2 | 6
  Psychological Abuse History | 6 | 8 | 14
Current contact with partner [Count of Participants; unit: Participants] | 28 | 26 | 54
Residence with target child before treatment [Count of Participants; unit: Participants] | 11 | 10 | 21
Physical violence toward coparent [Count of Participants; unit: Participants] | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Hostile Thoughts on the Articulated Thoughts in Simulated Situations Task
Description: Hostile Thinking coded from audio recorded transcripts. Participants are presented with 4 scenarios in which they are asked to respond verbally their thoughts about a given situation. The scenarios present incidents that could induce feelings of jealousy, anger, abandonment, or disrespect. These are coded for number of hostile cognitions by trained blind coders and summed for a total score. The range of scores is 0 to 28 . Higher scores mean greater hostile cognitions (worse outcome).
Time Frame: Baseline and intervention completion around 16 weeks
Population: Participants completed this assessment at baseline and 16 weeks only. We had some participants who refused to complete this specific measure at the post assessment and therefore we have less participants for analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Fathers for Change | Parent Education (PE)
Number analyzed (Participants) | 11 | 21
score on a scale
  Time 1-Baseline | 8.00 (1.90) | 7.62 (1.38)
  Time 2 - 16 weeks | 4.36 (1.43) | 4.23 (1.05)
Statistical Analysis 1: Comparison: Fathers for Change vs Parent Education (PE); Test type: Superiority; p > .10, Repeated Measures GLM; Time 2 at 16 weeks

2. Primary Outcome: Change in Total Score of the Difficulties With Emotion Regulation Scale (DERS)
Description: Emotion regulation difficulties are measured using this standardized self-report measure and a total score is calculated by summing the items. Score range is 0 to 180 with higher scores meaning worse outcome. Change over time is reported as the slope.
Time Frame: Baseline, intervention completion around 16 weeks, and 3 month post intervention around week 28
Measure: Mean (Standard Error); unit: ratio score baseline to 28 weeks
Arm/Group | Fathers for Change | Parent Education (PE)
Number analyzed (Participants) | 33 | 29
ratio score baseline to 28 weeks | -.31 (.13) | -.21 (.12)
Statistical Analysis 1: Comparison: Fathers for Change vs Parent Education (PE); Test type: Superiority; p < .01, GEE

3. Secondary Outcome: Change in Number of Domestic Violence Episodes on the Timeline Follow-Back Calendars
Description: Domestic Violence including physical and psychological aggression episodes across the length of followup. Higher scores mean more violence. Scores can range from 0 to 210 days. Change over time is reported as the slope.
Time Frame: Baseline through 3 month follow-up after intervention
Measure: Mean (Standard Deviation); unit: ratio score baseline to 28 weeks
Arm/Group | Fathers for Change | Parent Education (PE)
Number analyzed (Participants) | 33 | 29
ratio score baseline to 28 weeks | -.002 (.006) | -.01 (.007)
Statistical Analysis 1: Comparison: Fathers for Change vs Parent Education (PE); Test type: Superiority; p > .10, GEE

4. Secondary Outcome: Change in Total Score on the Adult Adolescent Parenting Inventory
Description: Overall score is indicator of maltreatment risk. A total score is calculated by summing the 5 scales with lower scores indicating greater risk for maltreatment. The range of scores is from 40 to 200. Change over time is reported as the slope.
Time Frame: Baseline, intervention completion around 16 weeks, and 3 month post intervention around week 28
Measure: Mean (Standard Error); unit: ratio score baseline to 28 weeks
Arm/Group | Fathers for Change | Parent Education (PE)
Number analyzed (Participants) | 33 | 29
ratio score baseline to 28 weeks | .12 (.07) | .03 (.07)
Statistical Analysis 1: Comparison: Fathers for Change vs Parent Education (PE); Test type: Superiority; p > .10, GEE

5. Secondary Outcome: Change in Coparenting Relationship Scale
Description: Brief Coparenting score which is calculated from a sum of 14 scale items. Scores range from 0 to 84 with higher scores indicating better coparenting. Change over time is reported as the slope.
Time Frame: Baseline, intervention completion around 16 weeks, and 3 month post intervention around week 28
Measure: Mean (Standard Error); unit: ratio score baseline to 28 weeks
Arm/Group | Fathers for Change | Parent Education (PE)
Number analyzed (Participants) | 33 | 29
ratio score baseline to 28 weeks | 0.06 (.11) | 0.02 (.08)
Statistical Analysis 1: Comparison: Fathers for Change vs Parent Education (PE); Test type: Superiority; p > .10, GEE

6. Secondary Outcome: Change in Days of Substance Use Reported on the Time Line Follow-Back Calendars
Description: Number of days of substance use over the course of the study. Higher scores equal more days of substance use. Possible range of scores was from 0 to 210 days. Change over time is reported as the slope.
Time Frame: At intervention completion (around week 16) and 3 months post intervention (at around 28 weeks)
Measure: Mean (Standard Error); unit: ratio score baseline to 28 weeks
Arm/Group | Fathers for Change | Parent Education (PE)
Number analyzed (Participants) | 33 | 29
ratio score baseline to 28 weeks | .01 (.01) | .03 (.03)
Statistical Analysis 1: Comparison: Fathers for Change vs Parent Education (PE); Test type: Superiority; p < .01, GEE

ADVERSE EVENTS:
Time Frame: Approximately 8 months
Arm/Group | Fathers for Change | Parent Education (PE)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/29
Serious Adverse Events (participants affected / at risk) | 2/33 | 0/29
Other Adverse Events (participants affected / at risk) | 10/33 | 5/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fathers for Change (N=33) | Parent Education (PE) (N=29)
Psychiatric hospitalization of child associated with study (Psychiatric disorders) | 1 (1) | 0 (0)
Child Protective Services Report (Investigations) | 1 (1) | 0 (0) — Father in the study reported child neglect of his children who were in the care of his step-father prompting a child protective services report.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fathers for Change (N=33) | Parent Education (PE) (N=29)
Participant Arrested and Jailed (Social circumstances) | 10 (10) | 5 (5) — Arrest due to probation violation, new drug charge or other reason resulting in jail time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT02979262/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT02979262/SAP_001.pdf